CLINICAL TRIAL: NCT06848114
Title: The Effect of Posture and Scapular Position on Performance Parameters in E-sport Players
Status: Completed | Type: Observational
Sponsor: Ömer Bayrak (Other)
Responsible Party: Sponsor-Investigator, Ömer Bayrak, Research Assistant, Halic University
Organization: Halic University (Other)
Other Study IDs: HUOBayrak
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Scapular Dyskinesis; Shoulder Proprioception; Reaction Time; Physical Activity; Posture; Hand-Eye Coordination
Keywords: Reaction time; Hand-eye coordination; Scapular dyskinesis; Posture; E-sport; Shoulder proprioception
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mobile E-sport Players: Mobile professional e-sports players compete at a high level within a team, participating in competitive mobile gaming.
- PC E-sport Players: PC professional e-sports players compete at a high level within a team, participating in competitive PC gaming.
- Control group: Individuals aged 18-25 years who played video games for less than 6 hours per week.

SUMMARY:
The research aims to examine how shoulder proprioception, scapular position, physical activity levels and posture influence key performance factors such as visual reaction time, audiotory reaction time and hand-eye coordination.

Various digital tools and tests will be utilized for assessment, including reaction time tests and hand-eye coordination evaluations conducted through HumanBenchmark and Audioreactiontime websites respectively, as well as posture analysis via mobile applications. Shoulder proprioception will be measured at specific flexion angles using a smartphone-based inclinometer, while scapular dyskinesis will be assessed through the lateral scapular sliding test. Additionally, participants' physical activity levels, assessed via the International Physical Activity Questionnaire (IPAQ), will be analyzed to determine potential correlations.

DETAILED DESCRIPTION:
E-sport is a competitive sport based on video games played professionally and multiplayer. To perform successfully in e-sport, high coordination and good reaction speed are essential. Studies indicate that prolonged inactivity and lack of physical activity in front of the computer can lead to weakening of motor skills and postural disorders. Additionally, abnormal positioning and movement of the scapula may reflect changes in the activity of surrounding muscles, potentially disrupting the coordinated movement with the humerus and possibly affect shoulder proprioception.

Based on this information, the investigators hypothesize that scapular dyskinesis and postural disorders in e-sport players affect their performance. The aim of our study is to investigate the impact of scapular position and posture on performance parameters, including hand-eye coordination, reaction time, shoulder proprioception, and physical activity among e-sport players.

For the assessment of visual reaction time, will be measured using the test on available on "humanbenchmark.com" will be used. Auditory reaction time will be measured using the test available on "playback.fm." Hand-eye coordination will be evaluated through the "Aim Reaction" test. Posture assessment will be conducted using the mobile application "PostureScreen."

Shoulder joint position sense will be assessed with the smartphone application "Clinometer" at 55°, 90°, and 125° shoulder flexion angles. Scapular dyskinesis will be evaluated using the lateral scapular sliding test at three different shoulder angles with a caliper.

The physical activity levels of the e-sport players will be determined using the International Physical Activity Questionnaire (IPAQ).

ELIGIBILITY:
Inclusion Criteria:

Individuals aged between 18 and 25 years. Professional engagement in PC or mobile e-sports for at least 6 hours per week continuously for the last six months.

PC professional e-sports players compete at a high level within a team, participating in competitive PC gaming.

Mobile professional e-sports players compete at a high level within a team, participating in competitive mobile gaming.

Control group: Individuals aged 18-25 years who played video games for less than 6 hours per week.

Exclusion Criteria For All Groups:

Any neurological, visual, or auditory impairment. History of upper extremity surgery. Use of medications known for their stimulant properties. Conditions that could interfere with test performance.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: E-sport Players in FUT E-sport Teams
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
The International Physical Activity Questionnaire (IPAQ) | Baseline
  The International Physical Activity Questionnaire (IPAQ) short form will assess e-sport players' physical activity levels. This validated questionnaire consists of seven items measuring time spent on walking, moderate, and vigorous activities, with energy expenditure expressed as MET minutes per week. The total score is calculated by summing the duration (minutes) and frequency (days) of each activity, while sedentary time is recorded separately. Only activities lasting at least 10 consecutive minutes are included.
  Scores are calculated as "MET minutes/week" by multiplying duration, frequency, and MET values: walking (3.3 METs), moderate (4 METs), and vigorous activity (8 METs). Physical activity levels are classified as:
  Physically inactive: <600 MET-min/week Low activity: 600-3000 MET-min/week Adequate activity: >3000 MET-min/week The Turkish IPAQ forms are validated for reliability.
Auditory Reaction Time Test | Baseline
  Auditory reaction time will be assessed using the playback.fm test (https://playback.fm/audio-reaction-time). Participants will press the "spacebar" on the keyboard upon hearing a sound. The test consists of five trials, and the average reaction time (ms) will be calculated from the recorded results.
Visual Reaction Time Test | Baseline
  Visual reaction time will be assessed using the "Reaction Time" test on the Human Benchmark website (https://humanbenchmark.com/tests/reactiontime). Participants will press a button as soon as the screen turns green. The test consists of five trials, and the average reaction time (ms) will be calculated from the recorded results.
Hand-Eye Coordination | Baseline
  The hand-eye coordination assessment is performed with the "Aim Reaction" test. The test is called "Aim Trainer" and is available on the website (https://humanbenchmark.com/tests/aim). At the beginning of the test, the participant tries to hit 30 targets on the screen as quickly and accurately as possible. After completing the test, the mean time to hit each target is displayed in milliseconds (ms)
Scapular Dyskinesis Assessment | Baseline
  Scapular dyskinesis will be assessed using a digital caliper based on the Kibler method, which has shown moderate to high reliability. The distance between the inferior angle of the scapula and the spinous process of the 7th thoracic vertebra (scapular distance) will be measured in centimeters (cm) across three positions:
  Arms at sides (0° abduction) Hands on iliac crest (45° abduction) 90° shoulder abduction with internal rotation Measurements are taken with the caliper's distal arm at the scapula's inferior angle and the proximal arm at the spinous process. Participants remain relaxed and focus on a fixed point. A ≥1.5 cm difference between scapulae indicates dyskinesis. The mean scapular distance is recorded for analysis.
Posture Assessment | Baseline
  Posture will be assessed using the mobile application "PostureScreen," employing the photographic method. The application calculates posture based on reference points marked on the anterior, posterior, and lateral aspects of a photograph. These reference points, along with athlete and assessor positioning, follow the guidelines outlined in the 2018 study by Iacob et al. The method is validated and reliable, with ICC scores ranging from 0.71 to 0.99.
  The application measures anterior and posterior shifts and tilts of the head, shoulders, chest, and hips, as well as lateral shifts and tilts of the head, shoulders, and hips. The total shift and tilt values are calculated as the sum of these measurements. These values will be used to generate a report detailing the participant's posture and its deviation from normal posture.
Shoulder Joint Position Sense | Baseline
  Shoulder joint position sense will be assessed using the "Clinometer" smartphone application (ICC = 0.98). The assessment follows a 5-minute warm-up with calisthenic exercises for the glenohumeral and scapulothoracic joints.
  The participant will be tested in shoulder flexion positions of 55°, 90°, and 125°. The smartphone is fixed between the shoulder and elbow to minimize deviations. The 55° position is first practiced with eyes open, then with eyes closed, holding for 10 seconds before returning to the starting position. The participant then identifies the target angle (55°) with eyes closed, responding with "OK" once reached. This process is repeated six times with 5-second rests between trials. Deviations from the target angle are recorded as absolute errors. The same procedure is followed for 90° and 125° flexion, for both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Haliç University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Werner BC, Holzgrefe RE, Griffin JW, Lyons ML, Cosgrove CT, Hart JM, Brockmeier SF. Validation of an innovative method of shoulder range-of-motion measurement using a smartphone clinometer application. J Shoulder Elbow Surg. 2014 Nov;23(11):e275-82. doi: 10.1016/j.jse.2014.02.030. Epub 2014 Jun 9. PMID 24925699
- [Background] Stewart HJ, Martinez JL, Perdew A, Green CS, Moore DR. Auditory cognition and perception of action video game players. Sci Rep. 2020 Sep 1;10(1):14410. doi: 10.1038/s41598-020-71235-z. PMID 32873819
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Keleş E, Şimşek E, Salmani M, Tarsuslu Şimşek T, Angın S, Yakut Y. (2016). Eklem hareket açıklığı ölçümünde kullanılan iki akıllı telefon uygulamasının uygulayıcı içi ve uygulayıcılar arası güvenirliğinin incelenmesi. J Exerc Ther Rehabil,3(1):21-29.
- [Background] Jenny, S. E., Manning, R. D., Keiper, M. C., Olrich, T. W. (2017). Virtual (ly) athletes: Where eSports fit within the definition of "sport". Quest, 69(1), 1-18.
- [Background] Hopkins, B. C. B. (2014). Validity of PostureScreen Mobile® in the measurement of standing posture.
- [Background] Hogan C, Corbett JA, Ashton S, Perraton L, Frame R, Dakic J. Scapular Dyskinesis Is Not an Isolated Risk Factor for Shoulder Injury in Athletes: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Aug;49(10):2843-2853. doi: 10.1177/0363546520968508. Epub 2020 Nov 19. PMID 33211975
- [Background] Hickey D, Solvig V, Cavalheri V, Harrold M, Mckenna L. Scapular dyskinesis increases the risk of future shoulder pain by 43% in asymptomatic athletes: a systematic review and meta-analysis. Br J Sports Med. 2018 Jan;52(2):102-110. doi: 10.1136/bjsports-2017-097559. Epub 2017 Jul 22. PMID 28735288
- [Background] Cretenoud AF, Barakat A, Milliet A, Choung OH, Bertamini M, Constantin C, Herzog MH. How do visual skills relate to action video game performance? J Vis. 2021 Jul 6;21(7):10. doi: 10.1167/jov.21.7.10. PMID 34269794
- [Background] Bloomer RJ, Martin KR, Pence JC. Impact of AmaTea(R) Max on physiological measures and gaming performance in active gamers: A placebo-controlled, double-blind, randomized study. J Clin Transl Res. 2022 Mar 1;8(2):93-102. eCollection 2022 Apr 29. PMID 35392125